CLINICAL TRIAL: NCT06473818
Title: Non-invasive vs Invasive Cardiac Output Monitoring in Patients Under Spinal Anesthesia During Cesarean Section: a Prospective Observational Study
Brief Title: Non-invasive vs Invasive Cardiac Output Monitoring During Cesarean Section
Status: Not yet recruiting | Type: Observational
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Yi Chen-2024-13
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Hemodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normotensive pregnant women: Singleton pregnancy ≥37 weeks, American Society of Anesthesiologists physical status classification I to II scheduled for cesarean section under spinal anesthesia
  Interventions: Device: Non-invasive monitoring; Device: Invasive monitoring

INTERVENTIONS:
Device: Non-invasive monitoring — Non-invasive cardiac output monitoring
  Other Names: Hemodynamics
Device: Invasive monitoring — Invasive cardiac output monitoring
  Other Names: hemodynamics

SUMMARY:
This study aims to evaluate the consistency of hemodynamic monitoring between NICAP and NICCO technologies (T20A; Chongqing, China) and the traditional pulse wave analysis method (EV1000; USA).

DETAILED DESCRIPTION:
The uterine placenta lacks autonomous regulatory ability, thus making maternal cardiac output (CO) the primary source of blood supply. Therefore, monitoring hemodynamics, including maternal CO, is of significant importance and provides guidance for anesthesia decisions such as fluid management and the administration of vasopressors during cesarean section. This study aims to evaluate the consistency of hemodynamic monitoring between NICAP and NICCO technologies (T20A; Chongqing, China) and the traditional pulse wave analysis method (EV1000; USA).

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years
* Primipara or multipara
* Singleton pregnancy ≥37 weeks
* American Society of Anesthesiologists physical status classification I to II
* Scheduled for cesarean section under spinal anesthesia

Exclusion Criteria:

* Body height < 150 cm
* Body weight > 100 kg or body mass index (BMI) ≥ 40 kg/m2
* Eclampsia or chronic hypertension or baseline blood pressure ≥140 mmHg
* Hemoglobin < 7g/dl
* Fetal distress, or known fetal developmental anomaly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Singleton pregnancy ≥37 weeks, American Society of Anesthesiologists physical status classification I to II scheduled for cesarean section under spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac output (CO) | 1-60 minutes after spinal anesthesia
  Monitoring data
Cardiac index (CI) | 1-60 minutes after spinal anesthesia
  Monitoring data
Stroke volume (SV) | 1-60 minutes after spinal anesthesia
  Monitoring data
Stroke volume variation (SVV) | 1-60 minutes after spinal anesthesia
  Monitoring data
Peripheral vascular resistance | 1-60 minutes after spinal anesthesia
  Monitoring data

SECONDARY OUTCOMES:
The incidence of post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia.
  Systolic blood pressure (SBP) < 80% of the baseline
The incidence of severe post-spinal anesthesia hypotension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) < 60% of the baseline
The incidence of bradycardia | 1-15 minutes after spinal anesthesia
  Heart rate < 60 beats/min
The incidence of nausea and vomiting. | 1-15 minutes after spinal anesthesia
  Presence of nausea and vomiting in patients after spinal anesthesia
The incidence of hypertension | 1-15 minutes after spinal anesthesia
  Systolic blood pressure (SBP) >120% of the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Yi Chen, M.D., Principal Investigator — General Hospital of Ningxia Medical University